CLINICAL TRIAL: NCT06491680
Title: Evaluation of the Cardioprotective Effect of Dapagliflozin on Anthracyclines-Induced Cardiotoxicity in Breast Cancer Patients
Brief Title: Cardiotoxicity in Breast Cancer Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Sara Mohamed Mohamed Abdel Motaleb, Lecturer of Clinical Pharmacy - Pharmacy Practice Department, Faculty of Pharmacy - Helwan University, Helwan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dapagliflozin
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: it is a randomized controlled trial for at least 40 breast cancer patients who receive 4 cycles of anthracyclines.
  These patients are divided into 2 groups . Group 1 take anthracyclines with dapagliflozin 10 mg and group 2 take anthracyclines only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin group (Active Comparator): Dapagliflozin group who consist of at least 20 breast cancer patients who receive 4 cycles of anthracyclines ( each cycle every 21 days ) with dapagliflozin 10 mg tablet once daily.
  Interventions: Drug: Dapagliflozin 10mg Tab
- Control group (No Intervention): Control group who consist of at least 20 breast cancer patients who receive 4 cycles of anthracyclines ( each cycle every 21 days ) only.

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin 10 mg tablet orally, once daily. Started 7 days before the first cycle of anthracyclines till the end of last anthracyclines dose.
  taken orally, once daily. Started from 5 to 7 days before the first cycle of anthracyclines till the end of last anthracycline dose.
  Other Names: Dapablix 10 mg
  Arms: Dapagliflozin group

SUMMARY:
The goal of this clinical trial is to learn if dapagliflozin drug has a cardioprotective effect against anthracyclines-induced cardiotoxicity. It will also learn about the safety of dapagliflozin drug.

Aim of the study:

Evaluate cardioprotective effect and safety of dapagliflozin against anthracyclines-induced cardiotoxicity.

The main questions it aims to answer are:

1. Does the drug lower the cardiotoxicity which induced by anthracyclines?
2. What medical problems do participants have when taking dapagliflozin drug?

Treatment

1. Anthracyclines by 4 cycles included doxorubicin 50-60 mg/m2 with cyclophosphamide 600 mg as a combination or epirubicin 90-100 mg/m2 with cyclophosphamide 600 mg as a combination.
2. Dapagliflozin 10 mg tablet orally, once daily. Started 7 days before the first cycle of anthracyclines till the end of last anthracyclines dose.

DETAILED DESCRIPTION:
Breast cancer is a malignant tumor that originates in the cells of the breast tissue. It is the most common cancer in women worldwide, accounting for 24.2% of all cancer cases among women.

According to the latest World Health Organization statistics, there were an estimated 2.3 million new cases of breast cancer in 2020; it is the second leading cause of cancer death in women after lung cancer.

In Egypt, breast cancer is the most common malignancy in women, accounting for 38.8% of cancers in this population, with the estimated number of breast cancer cases nearly 22,700 in 2022 and forecasted to be approximately 46,000 in 2050.

Anthracyclines are well-established and highly effective anti-neoplastic agents, used to treat several adult and pediatric cancers, such as breast cancer, leukemia, lymphomas, sarcomas, and many others.

Anthracycline-induced cardiotoxicity typically manifests as a reduction in left ventricular ejection fraction (LVEF), cardiomyopathy, or symptomatic congestive heart failure (CHF).

Acute anthracycline cardiotoxicity - occurs during or immediately after a single dose of an anthracycline. It may manifest as ventricular dysfunction, ECG abnormalities and arrhythmias.

Cardiotoxicity as a result of anthracycline chemotherapy has been linked to increased morbidity and mortality in breast cancer patients.

In a recently published cohort study, 2000 cancer survivors were monitored over 7 years. The authors found that approximately one-third of deaths could be attributed to long-term cardiotoxicity.

The specific mechanisms of anthracycline cardiotoxicity by Oxidative stress, which in the presence of iron, generates reactive oxygen species that cause lipid peroxidation of the cell membrane leading to damage of the cardiomyocytes, inflammation by up-regulating the levels of various inflammatory mediators, including interleukin-1 and tumor necrosis factor-α in the heart, subsequently leading to cardiomyocyte damage, In addition, DOX activated the nod-like receptor pyrin domain containing 3 (NLRP3) in cardiomyocytes, promoting cardiomyocyte apoptosis and down-regulation of sirtuin and adenosine monophosphate-activated protein kinase (AMPK) activity which associated with cardiovascular disease by enhanced apoptosis and increased fibrosis. The cardiomyocyte has always been considered the main cellular target of anthracycline toxic effect in the heart, as their destruction results in the progressive development of cardiac dysfunction.

Since anthracyclines is known to cause cardiotoxicity as a side effect, a baseline echocardiogram (ECHO) is ordered for each patient before initiating anthracycline chemotherapy treatment as a standard of care. Additionally, follow-up ECHOs are conducted after starting the treatment cycles to detect any early signs of cardiotoxicity.

Sodium Glucose co-transport inhibitors (SGLT2i) have demonstrated significant cardioprotective effects beyond their glucose-lowering capabilities. Recent clinical studies have highlighted their ability to reduce cardiovascular events, such as heart failure and myocardial infarction, in diabetic patients.

The cardioprotective benefits are thought to arise from multiple mechanisms, including improved cardiac energy metabolism, reduced blood pressure, and decreased fluid overload. As a result, SGLT2i are emerging as a crucial therapeutic option not only for glycemic control but also for enhancing heart health, marking a promising advancement in the management of cardiovascular risks.

SGLT2i significantly reduces Systolic Blood Pressure (SBP) and arterial stiffness that leads to better oxygen consumption by myocardium and hence lowers the cardiac afterload. It also helps in reducing the body weight slightly. Additionally, dapagliflozin also contributes by lowering the plasma volume by diuresis i.e., the increased excretion of sodium and glucose in urine. Decreasing the inflammation pathway by modulating the activation of NLRP3 inflammasome, thereby attenuating the synthesis of proinflammatory cytokines and reduced levels of tumor necrosis factor-α and interleukins, decreasing oxidative Stress by attenuate the generation of reactive oxygen species and enhance antioxidant mechanisms by inhibiting NADPH oxidase (nicotinamide adenine dinucleotide phosphate hydrogen ) and enhance energy metabolism by up-regulating the expression or activity of AMPK and sirtuins.

In light of the demonstrated cardioprotective effects of SGLT2 inhibitors (SGLT2i) in heart failure patients, these agents have been integrated into standard heart failure clinical guidelines, irrespective of the patient's diabetic status. Considering the well-established cardiotoxicity associated with anthracycline use, a thorough literature review was conducted to explore the potential of SGLT2i as adjunctive therapy to mitigate cardiac toxicity in breast cancer patients undergoing anthracycline-based chemotherapy. However, the search yielded only preclinical evidence, which highlighted the promising role of dapagliflozin. Consequently, this clinical trial aims to evaluate the efficacy of dapagliflozin as adjunctive therapy in breast cancer patients receiving anthracyclines, with a specific focus on preventing or delaying the onset of cardiotoxicity.

ELIGIBILITY:
Inclusion Criteria:

1. patients with pathologically proved invasive breast carcinoma.
2. Patients were indicated for anthracyclines containing adjuvant chemotherapy or new adjuvant anthracyclines.
3. Renal function (eGFR > 30 mL/minute per 1.73 m2 )
4. LVEF is more than 50 %
5. Age ≥ 18 and ≤ 60 years old

Exclusion Criteria:

1. patients with any cardiac condition that contraindicate the use of anthracyclines, like heart failure, arrythmia, stroke and myocardial infarction.
2. Previous anthracycline-containing regimens and any cardiotoxic chemotherapy regimens
3. pregnant or breastfeeding patients
4. patients receiving any other cardiotoxic agents.
5. Patients with diabetic ketoacidosis or patients with type 1 diabetes mellitus.
6. Mediastinal irradiation including heart.
7. Refusal to sign the written informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
N-terminal pro-B-type natriuretic peptide (NT-pro BNP) testing | Baseline and after the last cycle of anthracyclines ( 0 and 2 to 3 months from baseline)
  Monitoring the serum at Baseline and after the last cycle of anthracyclines. Changes in serum NT-Pro BNP from baseline will be calculated and compared between groups

SECONDARY OUTCOMES:
Echocardiography by measuring left ventricular ejection fraction (LVEF) | a) Baseline b) After the last cycle of anthracyclines (approximately 2 to 3 months from baseline) c) 3 months after the end of chemotherapy (approximately 5 to 6 months from baseline) d) As needed for any symptomatic patients
  LVEF (%) will be assessed using M-mode and 2D echocardiography performed by an experienced operator blinded to the patient's history. Changes in LVEF from baseline will be calculated and compared between groups at each time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Al demerdash hospital at oncology departement, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Dempke, Wolfram CM, et al. "Anthracycline-induced cardiotoxicity-are we about to clear this hurdle?." European Journal of Cancer 185 (2023): 94-104. — https://pubmed.ncbi.nlm.nih.gov/36966697/
- See also: Hwang, Hui-Jeong, et al. "Sodium-glucose cotransporter-2 inhibitors improve clinical outcomes in patients with type 2 diabetes mellitus undergoing anthracycline-containing chemotherapy: an emulated target trial. — https://www.nature.com/articles/s41598-023-48678-1
- See also: Kuo, Hsiao-Huai, et al. "Cardiovascular outcomes associated with SGLT2 inhibitor therapy in patients with type 2 diabetes mellitus and cancer: a systematic review and meta-analysis." Diabetology & Metabolic Syndrome 16.1 (2024): 108. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC11110336/
- See also: Henriksen, P, Rankin, S, Lang, N. Cardioprotection in Patients at High Risk of Anthracycline-Induced Cardiotoxicity: JACC: CardioOncology Primer. J Am Coll Cardiol CardioOnc. 2023 Jun, 5 (3) 292-297. — https://doi.org/10.1016/j.jaccao.2023.05.004
- See also: Dabour, Mohamed S., et al. "The Cardioprotective and Anticancer Effects of SGLT2 Inhibitors: JACC: CardioOncology State-of-the-Art Review." Cardio Oncology 6.2 (2024): 159-182. — https://doi.org/10.1016/j.jaccao.2024.01.007
- See also: Avagimyan, Ashot, et al. "Possibilities of dapagliflozin-induced cardioprotection on doxorubicin+ cyclophosphamide mode of chemotherapy-induced cardiomyopathy." International Journal of Cardiology 391 (2023): 131331. — https://doi.org/10.1016/j.ijcard.2023.131331